CLINICAL TRIAL: NCT00141986
Title: Pilot Trial of Vitamin D for the Prevention of Type 1 Diabetes
Brief Title: Feasibility Study of 2000 IU Per Day of Vitamin D for the Primary Prevention of Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Canadian Diabetes Association (Other)
Collaborators: Manitoba Medical Service Foundation (Other); Manitoba Institute of Child Health (Industry); The Health Sciences Centre Medical Staff Council (Unknown)
Responsible Party: Shayne P. Taback, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1622
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2005-09

CONDITIONS: Type 1 Diabetes
Keywords: vitamin D; type 1 diabetes; prevention trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D-higher dose (Experimental): Vitamin D 2000 IU per os once daily
  Interventions: Dietary Supplement: vitamin D3
- Vitamin D-lower dose (Active Comparator): Vitamin D 400 IU per os once daily
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3 — 2000 IU per day
  Other Names: cholecalciferol
  Arms: Vitamin D-higher dose
Dietary Supplement: vitamin D3 — 400 IU per os once daily
  Other Names: Cholecalciferol
  Arms: Vitamin D-lower dose

SUMMARY:
Type 1 diabetes is a common chronic disease of childhood. It is not yet preventable. Multiple daily injections of insulin, tests of blood sugar, and careful dietary planning are required lifelong to prevent long-term complications such as blindness and kidney failure. Recent studies of potential risk factors in children with diabetes, along with studies revealing the immunologic properties of vitamin D, and experiments in animals suggest higher doses of vitamin D may prevent type 1 diabetes. For proof for human children, a randomized trial will compare groups at risk randomly assigned to receive either the usual vitamin D supplement or a higher amount, 2000 IU daily. This initial study is a small scale test of procedures.

DETAILED DESCRIPTION:
Type 1 diabetes is a multifactorial disease with both strong genetic and non-genetic components of disease susceptibility. The uniquely strong genetic risk factor region, the human leukocyte antigen region on chromosome 6p, contributes approximately half of the genetic component and can be used for screening for diabetes risk. For example, individuals with the highest risk compound heterozygote genotype comprise 2% of the general population, but have a twenty fold increased risk for type 1 diabetes with an absolute risk of approximately 7% by age 15 years.

Studies of the non-inherited component of diabetes susceptibility implicate external environmental factors operating in the first year of life, suggesting the possibility to reverse the trend with the correct intervention. Recent data suggest that the vitamin D system is a potentially important target for therapeutic intervention to prevent type 1 diabetes. These data include epidemiological studies showing that vitamin D supplementation in infancy is associated with a substantially decreased subsequent risk of the disease, and animal work in the non-obese diabetes mouse model of autoimmune diabetes showing that the incidence of autoimmune diabetes increases when the animals are nutritionally deprived of vitamin D, and that the disease can be prevented using 1,25-dihydroxyvitamin D, and non-hypercalcemic vitamin D analogues. In vitro experiments suggest that the prevention seen in NOD mice may be due to combined effects of vitamin D on antigen presenting cells and activated T-cells.

Based on these epidemiological and animal model studies, we hypothesize that administration during infancy of cholecalciferol, the usual nutritional supplement form of vitamin D, at the increased dose of 2000 IU/day (instead of the current practice of 400 IU/day) will prevent type 1 diabetes in children from the general population at increased genetic risk.

The main objective of this proposal is to pilot a two-arm randomized controlled trial comparing these two doses. The participants are infants from the general population identified at increased genetic risk for type 1 diabetes by cord blood or filter paper blood spot HLA class II genetic screening. The study will measure key safety, compliance and pharmacokinetic, surrogate efficacy, and process outcomes including growth parameters, 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D levels, calcium levels in blood and urine, bone mineral content and body composition by densitometry, diabetes-related autoantibodies markers for beta-cell autoimmunity, and recruitment rates for both the screening and for the intervention trial.

ELIGIBILITY:
Inclusion Criteria:

* HLA genotypes that increase risk of type 1 diabetes: heterozygous for DRB1*03, DQA1*0501, DQB1*0201 / DRB1*04, DQA1*03011, DQB1*0302 (DRB1*04 ≠ *0403 or related alleles), or homozygous for DRB1*03, DQA1*0501, DQB1*0201, or homozygous for DRB1*04, DQA1*03011, DQB1*0302 (DRB1*04 ≠ *0403 or related alleles).

Exclusion Criteria:

* Premature, low birthweight, or major congenital malformations or serious chronic disease

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2003-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
change in 25(OH)D from baseline | at baseline (1 month of age), 2 months of age, 6 months of age, 9 months of age, 1 year of age
  25-hydroxyvitamin D levels

SECONDARY OUTCOMES:
renal ultrasound | 1 year of age
  to detect nephrocalcinosis
bone densitometry | at 6 months and 1 year of age
diabetes autoantibody levels | 1 year of age
  GADA, ICA-512, IAA
recruitment and retention rates | 1 year of age
Change from baseline in serum calcium levels | at baseline (1 month of age), 2 months of age, 6 months of age, 9 months of age, 1 year of age
changes in urine calcium:creatinine ratio | monthly in the first year of life

CONTACTS AND LOCATIONS:
Overall Officials: Shayne P Taback, MD FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- Manitoba Institute of Child Health, Winnipeg, Manitoba, Canada

REFERENCES:
- [Result] Wicklow BA, Taback SP. Feasibility of a type 1 diabetes primary prevention trial using 2000 IU vitamin D3 in infants from the general population with increased HLA-associated risk. Ann N Y Acad Sci. 2006 Oct;1079:310-2. doi: 10.1196/annals.1375.047. PMID 17130571